CLINICAL TRIAL: NCT03484026
Title: A Clinical Study of the Safety and Tolerability of BioFe, A Medical Food for the Management of Iron Deficiency
Brief Title: Safety and Tolerability of BioFe for Iron Deficiency Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidero Bioscience, LLC (Industry)
Collaborators: Milton S. Hershey Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 743376; 1R41DK105656-01A1 (NIH)
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Iron Deficiency
Keywords: Iron Deficiency; Anemia; Medical Food
MeSH Terms: conditions — Iron Deficiencies; Anemia

STUDY DESIGN:
Intervention Model Description: Consumption of BioFe in a single cohort of up to 8 subjects with iron deficiency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioFe Medical Food (Experimental): Consumption of BioFe Medical Food in a single cohort of up to 8 female subjects with iron deficiency.
  Interventions: Dietary Supplement: BioFe

INTERVENTIONS:
Dietary Supplement: BioFe — BioFe Medical Food is comprised of cultured nutritional/Baker's yeast (Saccharomyces cerevisiae) with high levels of Ferritin/Iron complex, pasteurized, and dried

SUMMARY:
This study evaluates the safety, tolerability, and activity of BioFe in the dietary management of iron deficiency in adults.

DETAILED DESCRIPTION:
Iron deficiency is the most common, widespread, and costly nutritional disorder worldwide with the World Health Organization (WHO) stating that up to 2 billion people are iron deficient. There is a serious and widespread misconception that oral iron supplements are safe and effective at alleviating iron deficiency. In a recent Cochrane review of 67 clinical trials, women taking oral iron supplements had a mere 38% decreased risk of iron deficiency compared to placebo. On the contrary, these subjects had a 114% increased risk of side effects, the vast majority of which were associated with gastrointestinal (GI) disturbance.

In infants and children, iron deficiency impedes mental, motor, and auditory neuronal development leading to serious lifelong cognitive and physical deficiencies. In adults, iron deficiency, and associated iron deficiency anemia, cause extreme fatigue, decreased immune system function and increased susceptibility to infectious disease, reduced work capacity, dizziness, headaches, hair loss, and generalized reduced quality of life. Iron deficiency is also linked to Restless Leg Syndrome (RLS), adult hearing deficits, reduced strength, coordination, and endurance, anxiety, increased heart failure morbidity, decreased intellectual performance, and erectile dysfunction among many others conditions.

Most iron deficient people are not effectively treated by, or are intolerant to, oral iron supplements. Intravenous iron repletion drugs effective, but are also costly and onerous to deliver leading to both patient and payor dissatisfaction.

BioFe, Medical Food for Iron Deficiency is nutritional/Baker's yeast (Saccharomyces cerevisiae), expressing the Ferritin protein. Ferritin is an indispensable iron storage, transport and absorption protein normally produced at low levels by almost all living organisms. An illustrative example of the biology of the Ferritin/Iron complex is its presence in human breast milk, providing infants the natural biological iron required for rapid learning and development, without gastrointestinal upset. BioFe provides high level expression of Ferritin that is naturally complexed with iron during culture, is pasteurized, and dried.

ELIGIBILITY:
Inclusion Criteria:

* Moderate iron deficiency defined as transferrin saturation (TSAT) <20% and serum ferritin <50 ng/mL.

Exclusion Criteria:

* Female subjects who are pregnant, plan to become pregnant, or not willing to use an acceptable form of contraception (tubal ligation or otherwise be incapable of pregnancy, hormonal contraceptives, spermicide plus barrier, or intrauterine device).
* Female subjects who are breastfeeding or plan to breastfeed after enrolling in the study.
* Hemochromatosis or other iron storage disorders.
* Hemoglobin below 8 g/dL.
* Previous gastric bypass, sleeve gastrectomy, or gastric band surgery.
* Currently on iron supplements and/or multivitamins containing iron (subjects may be pre-screened four weeks prior to the screening visit in order to stop/washout or switch to vitamins not containing iron).
* Currently on monoamine oxidase inhibitors (MAOIs) or Demerol.
* Current diagnosis of asthma and is actively using anti-asthmatic therapy.
* Smoking within two weeks of screening, current smoking, or anticipated smoking after enrolling in the study.
* Active malignancy within one year of screening.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than two times the upper limit of normal.
* Known positive Hepatitis B, Hepatitis C, or HIV-1/HIV-2.
* Unregulated hypertension, chronic kidney disease, irritable bowel syndrome, anemia of chronic diseases, chronic autoimmune inflammatory condition.
* Significant cardiovascular disease or congestive heart failure.
* Known allergy to yeast or any other component of BioFe.
* Received an investigational drug within 30 days of screening.
* Any laboratory abnormality, medical condition or psychiatric disorder, which in the opinion of the clinical principal investigator or Sponsor, may result in the subject being unable to comply with study requirements.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as the number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 18 Weeks
  Blood cell, blood chemistry, and stool sample analysis. Health questionnaires including GI symptoms, fatigue, and quality of life by the Short Form 36 (SF-36) questionnaire

SECONDARY OUTCOMES:
Correction of Iron Deficiency | 18 Weeks
  Increase in Serum Iron Measurements Ferritin, Iron, and TSAT

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wolfe, PhD, Study Chair — Sidero Bioscience, LLC; James R Connor, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Pennsylvania State University College of Medicine Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sidero Bioscience Website — http://www.siderobio.com/home.html